CLINICAL TRIAL: NCT04715620
Title: Efficacy and Safety of Niraparib Combined With Radiotherapy in Patients With Recurrent Glioblastoma
Brief Title: Niraparib Combined With Radiotherapy in rGBM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Jiang Wei, Professor, Tianjin Huanhu Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJHH-2306
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — niraparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- niraparib (Experimental)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib 300mg/day (body weight ≥77Kg and baseline platelet count ≥150,000/µL) or 200mg/day (body weight <77Kg or baseline platelet count <150,000/µL)

SUMMARY:
Thirty patients were enrolled in this study, mainly patients with first recurrence of glioblastoma, and the requirement is that they can receive secondary radiotherapy. Regardless of whether the patient has received a second operation or the MGMT promoter is methylated, they can be included in this study. After enrollment, patients were given niraparib 300mg/day (body weight ≥77Kg and baseline platelet count ≥150,000/µL) or 200mg/day (body weight <77Kg or baseline platelet count <150,000/µL), combined with radiotherapy (total dose 55Gy), follow-up Time 1 year. Until the patient has disease progression or intolerance or voluntarily withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* Sign a written informed consent form before conducting any research related procedures;
* Male or female aged between 18 and 70;
* Histologically confirmed WHO classification of recurrent glioblastoma grade IV;
* The expected survival time is more than 6 months
* Able to receive radiotherapy again
* KPS≥60
* Can swallow and maintain oral medication
* In the past month, no more than 3 grand epileptic seizures per week
* Good organ function, including: Bone marrow function: neutrophil count ≥1500/µL; platelets ≥100,000/µL; hemoglobin ≥10g/dL; Liver function: total bilirubin ≤1.5 times the upper limit of normal or direct bilirubin ≤1.0 times the upper limit of normal; AST and ALT ≤2.5 times the upper limit of normal; Renal function: serum creatinine ≤1.5 times the upper limit of normal value, or creatinine clearance ≥60mL/min (calculated according to Cockcroft-Gault formula);
* Ability to follow the plan;
* Any previous toxicity of chemotherapy has returned to ≤ CTCAE level 1 or baseline level, except for sensory neuropathy or alopecia with stable symptoms ≤ CTCAE level 2.

Exclusion Criteria:

* Those who are known to be allergic to niraparib or the active or inactive ingredients of drugs with similar chemical structure to niraparib;
* Those who have previously received PARP inhibitor therapy;
* Have received major surgery within 3 weeks before the start of the study, or any surgical effects that have not recovered after surgery or received chemotherapy;
* Received palliative radiotherapy with> 20% bone marrow 1 week before enrollment;
* The patient has previously or currently diagnosed myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
* Suffer from serious or uncontrolled diseases, including but not limited to:

Uncontrollable nausea and vomiting, inability to swallow study drugs, any gastrointestinal diseases that may interfere with drug absorption and metabolism; active viral infections such as human immunodeficiency virus, hepatitis B, hepatitis C, etc.; uncontrolled ventricular Arrhythmia, myocardial infarction in the last 3 months; uncontrolled grand mal seizures, unstable spinal cord compression, superior vena cava syndrome, or other mental disorders that affect the patient's informed consent; immunodeficiency (except splenectomy) Or other researchers believe that it may expose patients to high-risk toxic diseases; hypertension that cannot be controlled by drugs; and manifestations of intracranial hypertension, intracranial hemorrhage, and intracranial infarction caused by any reason;

* Patients with distant metastasis;
* Any past or current disease, treatment, or laboratory abnormality that may interfere with the results of the study, affect the patient's full participation in the study, or the investigator believes that the patient is not suitable for participating in the study; the patient must not be allowed within four weeks before the start of the study drug treatment Receive platelet or red blood cell transfusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
PFS-6 | 6 months
  6-month progression-free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, Principal Investigator — Tianjin Huanhu Hospital
Locations (1):
- Tianjin Huanhu Hosptal, Tianjin, Tianjin Municipality, China